CLINICAL TRIAL: NCT00746356
Title: A Clinical Evaluation of the Current™ Radio Frequency (RF) Implantable Cardioverter Defibrillator (ICD) Models 2215/1215 and Promote™ RF Cardiac Resynchronization Therapy Defibrillator (CRT-D) Model 3215 Pulse Generators
Brief Title: Safety and Efficacy of Automatic Testing Feature in New ICDs and CRT-Ds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 40005027; IDE # G080060 (Other: FDA); Doc number 40005027 (Other: St. Jude Medical)
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Results first posted 2013-03-01 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure; Ventricular Arrythmias
Keywords: heart failure; cardiac resynchronization therapy; autocapture; Current RF; Promote RF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Promote RF CRT-D (Experimental): Patients with CRT-D device will have the autocapture features of the device tested.
  Interventions: Device: Testing of the autocapture features of the device
- Current RF ICD (Experimental): Patients with ICD device will have the autocapture features of the device tested.
  Interventions: Device: Testing of the autocapture features of the device

INTERVENTIONS:
Device: Testing of the autocapture features of the device — Patients receiving cardiac resynchronization therapy will have new autocapture features tested on right atrial, right ventricular and left ventricular leads.
  Arms: Promote RF CRT-D
Device: Testing of the autocapture features of the device — Patients with an Implantable Cardioverter Defibrillator will have new autocapture features tested on the right atrial and right ventricular leads.
  Arms: Current RF ICD

SUMMARY:
This study is a prospective, non-randomized, multi-center clinical trial that will assess the safety and effectiveness of investigational models of the Promote™ RF CRT-D and Current™ RF ICD devices. These new ICD and CRT-D devices have new features that allow the device to periodically check how much energy is needed to pace a patient's heart and to automatically adjust the amount of energy used to pace the heart.

DETAILED DESCRIPTION:
All patients enrolled in the study will have their device tested to determine if the device can automatically measure how much energy is needed to pace the patient's heart. If the test is successful, the patient's device will be programmed to turn that feature on. 3 months after enrollment, the patient will return to the clinic to have their device re-tested using an automatic test method to measure the amount of energy needed to make the patient's heart beat. A manual test method will also be used to measure the amount of energy needed to make the patient's heart beat. The intent of the study is to show the automatic method works just as well as the manual method.

ELIGIBILITY:
Inclusion Criteria:

* Have an approved indication, as outlined by American Heart Association/Heart Rhythm Society (AHA/HRS) guidelines, for implantation of an ICD or CRT-D for the treatment of life-threatening ventricular tachyarrhythmia(s) or heart failure, or undergo revision of their ICD or CRT-D system to replace the pulse generator.
* Have the ability to provide informed consent for study participation and be willing and able to comply with the prescribed follow-up tests and schedule of evaluations.

Exclusion Criteria:

* Have a classification of Status 1 for cardiac transplantation or consideration for transplantation over the next 3 months.
* Have had a recent myocardial infarction, unstable angina or cardiac revascularization (percutaneous transluminal coronary angioplasty (PTCA), Stent or Coronary Artery Bypass Graft(CABG)) within 40 days of enrollment.
* Have had a recent cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 3 months of enrollment.
* Are allergic to dexamethasone sodium phosphate (DSP).
* Be currently participating in a clinical investigation that includes an active treatment arm.
* Be pregnant or are planning for pregnancy within 6 months following enrollment.
* Have a life expectancy of less than 6 months.
* Be less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Shipman, Study Director — Director, Clinical Affairs, St. Jude Medical
Locations (5):
- United States (5):
  - Arkanasas Heart Hospital, Little Rock, Arkansas
  - Baptist Health Hospital, Little Rock, Arkansas
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - St. Thomas Hospital, Nashville, Tennessee
  - Southwest Texas Methodist Hospital, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in August 2008 at hospitals where patients were being implanted with implantable cardioverter defibrillators or in and physician offices where these patients were being followed. Recruitment was completed on April 1, 2009.
Pre-assignment Details: All patients who were enrolled in the study had the autocapture feature tested at each study visit, starting with at the implant visit when the study device was implanted.
Groups:
- CRT-D Device Patients: All patients with a cardiac resynchronization therapy device (CRT-D)enrolled in the study.
- ICD Device Patients: All patients with an implantable cardioverter defibrillator (ICD) device enrolled in the study.
Period: Overall Study
Arm/Group | CRT-D Device Patients | ICD Device Patients
Started | 81 | 47
Completed | 70 | 40
Not Completed | 11 | 7
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Death | 7 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Removal of Device | 0 | 1
Not completed — Patient relocated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All patients enrolled in the study
Arm/Group | All Patients
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 96
Cardiomyopathy [Number; unit: Participants]
  Ischemic Etiology | 87
  Non-Ischemic Etiology | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Free of System-related Complications at 3-months Post Implant
Time Frame: 3 months post implant
Measure: Number; unit: Percentage of Participants
Groups:
- Participants Successfully Implanted With Devices: All participants successfully implanted with an ICD or CRT-D
Arm/Group | Participants Successfully Implanted With Devices
Number analyzed (Participants) | 128
Percentage of Participants | 93.6 [lower limit 89.9]

2. Primary Outcome: Atrial AutoCapture (ACap) Confirm Effectiveness Endpoint - Absolute Difference Between the Automatic and Manual Capture Threshold Test
Description: Atrial AutoCapture Confirm is an automatic test that the device performs without any interaction by the physician and is one of the features being evaluated in the study. The test temporarily decreases the atrial pacing voltage until it determines that the device is no longer capturing the atria. That value is reported to the physician when the device is read by the programmer. This endpoint looks at the absolute difference between this automated test and a manual test in which the physician decreases the atrial pulse voltage and determines the atrial threshold by viewing the EKG.
Time Frame: 3 months post implant
Population: Per protocol, the first 19 participants who successfully completed both an automatic and manual capture threshold test were included in this analysis.
Measure: Mean (Standard Deviation); unit: Volts
Groups:
- Participants With Dual Chamber ICDs or CRTD Devices: Per protocol, the first 19 participants who successfully completed both an automatic and manual capture threshold
Arm/Group | Participants With Dual Chamber ICDs or CRTD Devices
Number analyzed (Participants) | 19
Volts
  Atrial AutoCapture Threshold | 0.743 (0.357)
  Manual Capture Threshold | 0.737 (0.195)
Statistical Analysis 1: Comparison: Participants With Dual Chamber ICDs or CRTD Devices; The null hypothesis was rejected at significance level 1.67% if the mean difference between the automatic test and the manual test was <0.25 volts; Test type: Non-Inferiority or Equivalence — Sample size was calculated for an 80% power to reject the null hypothesis at 1.67% significance level; p < 0.0001, t-test, 1 sided — P-value was adjusted for multiple efficacy endpoints. If all three primary effectiveness endpoints were met a value of 5% was used, if two were met a value of 2.5% was used, and if one was met a value of 1.67% was used; If the data is not normally distributed, then the Wilcoxon signed rank test will be used to perform the two one-sided testing; Mean Difference (Final Values) = 0.0066, 95% CI 1-sided [lower limit -0.25], Standard Deviation 0.3103

3. Primary Outcome: Ventricular Autocapture Effectiveness Endpoint - Absolute Difference Between the Automatic and Manual Capture Threshold Test
Description: Ventricular AutoCapture is an automatic test that the device performs without any interaction by the physician and is one of the features being evaluated in the study. The test temporarily decreases the ventricular pacing voltage until it determines that the device is no longer capturing the ventricles. That value is reported to the physician when the device is read by the programmer. This endpoint looks at the absolute difference between this automated test and a manual test in which the physician decreases the ventricular pulse voltage and determines the ventricular threshold by viewing the EKG.
Time Frame: 3 months post implant
Population: Per protocol, the first 38 participants with an ICD who successfully completed both an automatic and manual capture threshold test were included in this analysis.
Measure: Mean (Standard Deviation); unit: Volts
Groups:
- Participants With Single or Dual Chamber ICDs: Per protocol, the first 38 participants with an ICD who successfully completed both an automatic and manual capture threshold in the right ventricle
Arm/Group | Participants With Single or Dual Chamber ICDs
Number analyzed (Participants) | 38
Volts
  Automatic Capture Threshold | 0.809 (0.405)
  Manual Capture Threshold | 0.862 (0.442)
Statistical Analysis 1: Comparison: Participants With Single or Dual Chamber ICDs; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size was calculated for an 80% power to reject the null hypothesis at 1.67% significance level; p = 0.0001, t-test, 1 sided — P-value was adjusted for multiple efficacy endpoints. If all three primary effectiveness endpoints were met a value of 5% was used, if two were met a value of 2.5% was used and if one was met a value of 1.67% was used; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.0625, 95% CI 1-sided [lower limit -0.25], Standard Deviation 0.0948

4. Primary Outcome: Right Ventricular (RV) AutoCapture Effectiveness Endpoint - Difference Between the Automatic and Manual Capture Threshold Test
Description: Right Ventricular AutoCapture is an automatic test that the device performs without any interaction by the physician and is one of the features being evaluated in the study. The test temporarily decreases the ventricular pacing voltage until it determines that the device is no longer capturing the ventricles. That value is reported to the physician when the device is read by the programmer. This endpoint looks at the absolute difference between this automated test and a manual test in which the physician decreases the ventricular pulse voltage and determines the ventricular threshold by viewing the EKG.
Time Frame: 3 months post implant
Population: Per protocol, the first 43 CRT-D participants who successfully completed both an automatic and manual capture threshold in the right ventricle were included in this analysis.
Measure: Mean (Standard Deviation); unit: Volts
Groups:
- Participants With CRT-D Devices: Per protocol, the first 43 CRT-D participants who successfully completed both an automatic and manual capture threshold in the right ventricle
Arm/Group | Participants With CRT-D Devices
Number analyzed (Participants) | 43
Volts
  Automatic Capture Threshold | 0.739 (0.279)
  Manual Capture Threshold | 0.794 (0.278)
Statistical Analysis 1: Comparison: Participants With CRT-D Devices; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size was calculated for an 80% power to reject the null hypothesis at 1.67% significance level; p = 0.0001, t-test, 1 sided — P-value was adjusted for multiple efficacy endpoints. If all three primary effectiveness endpoints were met a value of 5% was used, if two were met, a value of 2.5% were used and if one was met a value of 1.67% was used; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.0556, 95% CI 1-sided [lower limit -0.25], Standard Deviation 0.0824

5. Primary Outcome: Left Ventricular (LV) AutoCapture Effectiveness Endpoint - Difference Between the Automatic and Manual Capture Threshold Test
Description: Left Ventricular AutoCapture is an automatic test that the device performs without any interaction by the physician and is one of the features being evaluated in the study. The test temporarily decreases the ventricular pacing voltage until it determines that the device is no longer capturing the ventricles. That value is reported to the physician when the device is read by the programmer. This endpoint looks at the absolute difference between this automated test and a manual test in which the physician decreases the ventricular pulse voltage and determines the ventricular threshold by viewing the EKG.
Time Frame: 3 months post implant
Population: Per protocol, the first 43 CRT-D participants who successfully completed both an automatic and manual threshold in the left ventricle were included in the analysis.
Measure: Mean (Standard Deviation); unit: Volts
Groups:
- Participants With CRT-D Devices: Per protocol, the first 43 CRT-D participants who successfully completed both an automatic and manual threshold in the left ventricle.
Arm/Group | Participants With CRT-D Devices
Number analyzed (Participants) | 43
Volts
  Automatic Capture Threshold | 1.458 (0.631)
  Manual Capture Threshold | 1.456 (0.618)
Statistical Analysis 1: Comparison: Participants With CRT-D Devices; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size was calculated for an 80% power to reject the null hypothesis at 1.67% significance level; p = 0.0001, t-test, 1 sided — P-value was adjusted for multiple efficacy endpoints. If three primary effectiveness endpoints were met a value of 5% was used, if two were met a value of 2.5% was used and if one was met a value of 1.67% was used; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.0028, 95% CI 1-sided [lower limit -0.25], Standard Deviation 0.2852

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/128
Other Adverse Events (participants affected / at risk) | 33/128
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=128)
ecchymosis at implant site (Surgical and medical procedures) | 1 (1) — Adverse events are reported as either a complication or observation (1), defined as an adverse event that requires invasive intervention or an adverse event that can be managed without invasive intervention, respectively.
hematoma (Surgical and medical procedures) | 7 (7) — 7 observations
LV lead dislodgement (Surgical and medical procedures) | 1 (1) — 1 complication
pericardial tamponade (Surgical and medical procedures) | 1 (1) — 1 complication
erroneous elective replacement alert (Surgical and medical procedures) | 3 (3) — 3 observations
high defibrillation thresholds (Cardiac disorders) | 1 (1) — 1 observation
infection (Surgical and medical procedures) | 2 (2) — 1 complication, 1 observation
suspected set screw malfunction (Surgical and medical procedures) | 1 (1) — 1 complication
suspected generator malfunction (Surgical and medical procedures) | 1 (1) — 1 complication
elevated pacing thresholds - RA lead (Cardiac disorders) | 1 (1) — 1 observation
elevated pacing thresholds - RV lead (Cardiac disorders) | 2 (2) — 1 complication, 1 observation
elevated pacing threshold - LV lead (Cardiac disorders) | 9 (9) — 9 observations, 9 pts
lead dislodgement/migration - RA lead (Surgical and medical procedures) | 2 (2) — 2 complications - 2 pts
lead dislodgement/migration - RV lead (Surgical and medical procedures) | 1 (1) — 1 complication
lead dislodgement/migration - LV lead (Surgical and medical procedures) | 3 (4) — 4 complications, 3 pts
lead insulation damage - RV lead (Surgical and medical procedures) | 1 (1) — 1 complication
phrenic nerve/diaphragmatic stimulation - LV lead (Surgical and medical procedures) | 5 (5) — 4 observations, 1 complication
RA and RV lead dislodgement/migration (Surgical and medical procedures) | 1 (1) — 1 observation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less